CLINICAL TRIAL: NCT00964275
Title: Study of Positron Emission Tomography With 18-fluorodeoxyglucose in Detecting Cancer in Patients With Idiopathic Venous Thromboembolism
Brief Title: Standard Diagnostic Procedures With or Without Fludeoxyglucose F 18 Positron Emission Tomography in Finding Cancer in Patients With a Blood Clot in a Vein
Acronym: MVTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000639720; HCB-MVTEP; RB 08-062; INCA-RECF0945; EUDRACT-2008-004135-38
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Thromboembolism; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo diagnostic fludeoxyglucose F 18 PET in addition to standard methods.
  Interventions: Radiation: fludeoxyglucose F 18
- Arm II (Active Comparator): Patients only undergo standard diagnostic methods.
  Interventions: Procedure: diagnostic procedure

INTERVENTIONS:
Procedure: diagnostic procedure — Standard diagnostic procedures followed
  Arms: Arm II
Radiation: fludeoxyglucose F 18 — PET with flueoxyglucose F 18
  Arms: Arm I

SUMMARY:
RATIONALE: Diagnostic procedures, such as fludeoxyglucose F 18 positron emission tomography, may help find and diagnose cancer. It is not yet known whether standard diagnostic procedures are more effective when given with or without fludeoxyglucose F 18 positron emission tomography in finding cancer.

PURPOSE: This randomized clinical trial is studying fludeoxyglucose F 18 positron emission tomography given together with standard diagnostic procedures to see how well it works compared with standard diagnostic procedures alone in finding cancer in patients with a blood clot in a vein.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Demonstrate the efficacy, in terms of increased numbers of cancer diagnoses, of PET-CT with 18-FDG in patients with idiopathic venous thromboembolism.

Secondary

* Assess the risk of cancer detected at 1 year.
* Assess whether PET allows earlier detection of cancer.
* Evaluate survival.

OUTLINE: This is a multicenter study.

All patients undergo standard (clinical and biological) diagnostic tests for cancer. Patients are randomized to 1 of 2 diagnostic arms.

* Arm I: Patients undergo diagnostic fludeoxyglucose F 18 PET in addition to standard methods.
* Arm II: Patients only undergo standard diagnostic methods. Patients are followed up for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of idiopathic venous thromboembolism (IVTE) meeting 1 of the following criteria:

  * Newly diagnosed
  * Recurrent disease controlled by anticoagulant therapy
* No IVTE caused by a reversible major risk factor
* No IVTE caused by a major constitutional risk factor, including any of the following:

  * Antiphospholipid antibody syndrome
  * Antithrombin deficit
  * Protein C
  * Protein S

PATIENT CHARACTERISTICS:

* Not pregnant
* No other known active cancer at the onset of IVTE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of cancers diagnosed | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Salaun, MD, Principal Investigator — CHU Brest - Hopital De La Cavale Blanche
Locations (1):
- CHU Brest - Hopital De La Cavale Blanche, Brest, France

REFERENCES:
- [Derived] Robertson L, Broderick C, Yeoh SE, Stansby G. Effect of testing for cancer on cancer- or venous thromboembolism (VTE)-related mortality and morbidity in people with unprovoked VTE. Cochrane Database Syst Rev. 2021 Oct 1;10(10):CD010837. doi: 10.1002/14651858.CD010837.pub5. PMID 34597414
- [Derived] Robin P, Le Roux PY, Tromeur C, Planquette B, Prevot-Bitot N, Lavigne C, Pastre J, Merah A, Couturaud F, Le Gal G, Salaun PY. Risk factors of occult malignancy in patients with unprovoked venous thromboembolism. Thromb Res. 2017 Nov;159:48-51. doi: 10.1016/j.thromres.2017.08.021. Epub 2017 Sep 28. PMID 28978463
- [Derived] Robin P, Le Roux PY, Planquette B, Accassat S, Roy PM, Couturaud F, Ghazzar N, Prevot-Bitot N, Couturier O, Delluc A, Sanchez O, Tardy B, Le Gal G, Salaun PY; MVTEP study group. Limited screening with versus without (18)F-fluorodeoxyglucose PET/CT for occult malignancy in unprovoked venous thromboembolism: an open-label randomised controlled trial. Lancet Oncol. 2016 Feb;17(2):193-199. doi: 10.1016/S1470-2045(15)00480-5. Epub 2015 Dec 8. PMID 26672686